CLINICAL TRIAL: NCT00965510
Title: Improved Management of Type II Diabetes in a Primary Care Office With Targeted Case Management
Brief Title: SeaCare's Care Coordination for Diabetes Management in a Primary Care Office
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment of control and study patients
Sponsor: SeaCare Health Services (Other)
Collaborators: New Hampshire Charitable Foundation (Unknown)
Responsible Party: Gwendolyn Gladstone, MD, SeaCare Health Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9118277Downing306
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Type 2 Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care Coordination (Experimental): Patients receive care coordination to improve their diabetes.
  Interventions: Behavioral: care coordination
- control (No Intervention): patients with type II diabetes receive usual health care

INTERVENTIONS:
Behavioral: care coordination — patients receive care coordination to improve their type II diabetes
  Arms: Care Coordination

SUMMARY:
The purpose of this study is to determine whether it is possible to improve health outcomes for patients with Type II diabetes, a community-based health care agency will offer care coordination to half of a study group in a family practice office. The intervention will include assessing patients' status using two instruments:

a depression screen (the PHQ9) and a motivation to change scale (the Patient Activation Measure, PAM). A masters-level social worker will counsel patients in the intervention group. Changes in patients' health status, PHQ9 scores and PAM scores over one year will be measured. Outcomes will be compared between the study group and the group without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type II

Exclusion Criteria:

* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Scores on PHQ9, PAM and health indicators | 1 year

SECONDARY OUTCOMES:
Satisfaction with care coordination model. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Gladstone, MD, Principal Investigator — SeaCare Health Services
Locations (1):
- Exeter Family Care, Exeter, New Hampshire, United States